CLINICAL TRIAL: NCT05656261
Title: APOL1 Genetic Testing in African Americans: Exploring Attitudes About Genetic Risk to Improve Comprehensive Kidney Risk Assessment for Patients and Families
Brief Title: APOL1 Genetic Testing in African Americans
Status: Recruiting | Type: Observational
Sponsor: St. Louis University (Other)
Collaborators: Mid-America Transplant (Other)
Responsible Party: Principal Investigator, Krista Lentine MD, PhD, Principal Investigator, St. Louis University
Other Study IDs: 29188
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Genetic Predisposition; Chronic Kidney Diseases; Nephropathy; APOL1 Associated Kidney Disease; Disparities
Keywords: APOL1 Renal Risk Variants
MeSH Terms: conditions — Genetic Predisposition to Disease; Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will have the option to consent or decline to have their remaining blood sample biobanked and stored to be used for future research studies. All samples and data approved for future research will be deidentified to protect patient confidentiality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults of African or sub-Saharan ancestry: The study focuses on those who are at risk of having the APOL1 renal risk variants, which homozygous or compound heterozygous variants have been shown to lead to Chronic Kidney Disease in some of the population. Those who are found to have this mutations are of African or sub-Saharan ancestry. This study will include those aged 18-90 of this population.
  Interventions: Genetic: Assessment of the frequency of APOL-1 renal risk variant in the black population, and evaluating their attitudes about genetic testing and APOL1 genotype via self-administered surveys

INTERVENTIONS:
Genetic: Assessment of the frequency of APOL-1 renal risk variant in the black population, and evaluating their attitudes about genetic testing and APOL1 genotype via self-administered surveys — On day of enrollment, participants will have 1 blood sample obtained to extract DNA for determining their APOL1 genotype, and will answer a survey asking about their attitudes/beliefs on kidney disease, hypertension, and diabetes, as well as genetic testing. Participants will receive their results via telephone shortly thereafter, and then complete the same survey at 3 months and 12 months post-enrollment, in order to evaluate if any of their attitudes or beliefs have changed since knowing their APOL1 genetic test result. Those who are interested, specifically those who carry the homozygous or compound heterozygous renal risk variant, will have the option to speak with a designated genetic counselor who is associated with the study site and approved by the IRB.

SUMMARY:
Recent breakthroughs in medical genetics have discovered that a portion of kidney failure affecting the Black community is mediated by coding variants in a gene called apolipoprotein L1 (APOL1) - and that genetic variants, not race - account for increased risk. For APOL1 genetic testing to be applied in a manner that improves patient care and outcomes, more information is needed regarding associations of genotype with clinical parameters related to kidney health. Further, understanding patient perceptions about knowledge of the results of APOL1 genetic testing, and how that impacts patient engagement with management of hypertension and other renal risk factors, is urgently needed.

* In a Phase 1 pilot study, we offered APOL1 genetic testing to Black patients seen in our Hypertension and Nephrology clinics at Saint Louis University, an academic medical center that serves the local urban community, and surveyed patients on attitudes and concerns about APOL1 genetic testing. 144 participants were enrolled in Phase 1.
* In the Phase 2 study, we will advance this important work in our community by offering participation to a broader patient base, including patients seen in Internal and Family Medicine clinics, SLU Hospital, as well as to first-degree relatives and spouses of SLUCare participants. This expansion seeks to advance understanding of environment-gene interactions, improve risk prediction, and target management of potentially modifiable risk factors.

DETAILED DESCRIPTION:
Recent recognition of coding variants in the Apolipoprotein L1 (APOL1) gene as a strong risk factor for advanced chronic kidney disease (CKD) and end-stage kidney disease (ESKD) in African Americans (AAs) has marked one of the most impactful discoveries in kidney precision medicine. It is well-established that AAs have an increased risk of kidney failure, but it now appears that at least a portion of this risk disparity is genetically mediated by APOL1 renal risk variants (RRVs). Approximately 13% of Black Americans have APOL1 high-risk genotypes (2 copies of G1, G2, or compound heterozygotes [2 RRVs]) and are at higher risk for ESKD. Importantly, APOL1 high-risk genotypes are not deterministic for kidney disease. Rather, additional genetic and/or environmental "second hits" are likely required for disease initiation and progression. These "second hits" may include environmental factors and social determinants of health, as well as biologic factors.

Supported by the Mid-America Transplant Foundation, this study seeks to assess the frequency of APOL1 RRVs in local African American patients with hypertension and to assess their attitudes about APOL1 genetic testing and the potential impact of knowing one's APOL1 genotype on hypertension and renal risk factor management through self-administered surveys.

This study is open to Black patients seen in SLUCare Nephrology, Hypertension, Internal/Family Medicine clinics, or the University hospital, as well as to first-degree relatives and household family members (e.g. spouses) of enrolled participants or previously APOL1 genotyped patients of SSM Saint Louis University Hospital and SLUCare clinic. Family-based recruitment may help discriminate impacts of genetic risk from other potential shared biologic and non-biologic risk factors, and will also broaden the reach of the project in our community.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-90
* Self-Identified as Black/African American. Race will be self-identified. Patients of African ancestry who identify as multi-racial are also eligible to participate.

Exclusion Criteria:

* Cognitively impaired/unable to provide consent
* Terminally ill
* Renal replacement therapy (RRT), e.g., (but not limited to) hemodialysis, peritoneal dialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Black patients seen at Saint Louis University Internal Medicine, Family Medicine, Hypertension and Nephrology Clinics
  * Family members on enrolled patients, including first-degree relatives and household family members (e.g. spouses). Up to 3 family members per enrolled patient may also be enrolled.
  * Participation is also open to family members of SLUCare patients who have undergone APOL1 genotyping as part of clinical care (i.e., during evaluation of chronic kidney disease, including for kidney transplantation evaluation, or during living donor candidacy evaluation)
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine frequency of APOL1 renal risk variants in black population | 1 year
  To assess the frequency and sociodemographic/clinical correlates of APOL1 renal risk variants in a local urban population of Black patients seen in Nephrology, Hypertension, Internal/Family Medicine clinics, or University Hospital.

SECONDARY OUTCOMES:
Determine frequency of first degree relatives of enrolled participants with APOL1 renal risk variants | 1 year
  To assess the association and interaction between potential "second hits" such as environmental factors and comorbidities with APOL1 genotype on kidney function among Black patients and their families.
  * To assess attitudes of patients and family members about APOL1 genetic testing and the potential impact of knowing one's APOL1 genotype on hypertension and renal risk factor management through self-administered surveys.
  * To assess the interest of patients and family members in genetic counseling related to APOL1 genetic testing and kidney risk.

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Health Saint Louis University Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lentine KL, Muiru AN, Lindsay KK, Caliskan Y, Edwards JC, Memon AA, Mosman AK, Miyata KN, Vo TM, Freedman BI, Carriker A, Hsu CY, Philipneri MD. APOL1 Genetic Testing in Patients With Recent African Ancestry and Hypertension: A Pilot Study of Attitudes and Perceptions. Kidney Med. 2022 Sep 29;4(12):100549. doi: 10.1016/j.xkme.2022.100549. eCollection 2022 Dec. No abstract available. PMID 36573119
- [Result] Genovese G, Friedman DJ, Ross MD, Lecordier L, Uzureau P, Freedman BI, Bowden DW, Langefeld CD, Oleksyk TK, Uscinski Knob AL, Bernhardy AJ, Hicks PJ, Nelson GW, Vanhollebeke B, Winkler CA, Kopp JB, Pays E, Pollak MR. Association of trypanolytic ApoL1 variants with kidney disease in African Americans. Science. 2010 Aug 13;329(5993):841-5. doi: 10.1126/science.1193032. Epub 2010 Jul 15. PMID 20647424
- [Result] Friedman DJ, Kozlitina J, Genovese G, Jog P, Pollak MR. Population-based risk assessment of APOL1 on renal disease. J Am Soc Nephrol. 2011 Nov;22(11):2098-105. doi: 10.1681/ASN.2011050519. Epub 2011 Oct 13. PMID 21997396
- [Result] Anyaegbu EI, Shaw AS, Hruska KA, Jain S. Clinical phenotype of APOL1 nephropathy in young relatives of patients with end-stage renal disease. Pediatr Nephrol. 2015 Jun;30(6):983-9. doi: 10.1007/s00467-014-3031-0. Epub 2014 Dec 23. PMID 25530085
- [Result] Freedman BI, Langefeld CD, Turner J, Nunez M, High KP, Spainhour M, Hicks PJ, Bowden DW, Reeves-Daniel AM, Murea M, Rocco MV, Divers J. Association of APOL1 variants with mild kidney disease in the first-degree relatives of African American patients with non-diabetic end-stage renal disease. Kidney Int. 2012 Oct;82(7):805-11. doi: 10.1038/ki.2012.217. Epub 2012 Jun 13. PMID 22695330
- [Derived] Abu Al Rub F, Elsurer Afsar R, Fleetwood VA, Bastani B, Randall H, Nazzal M, Varma C, Afsar B, Jackson H, Yount S, Wooley C, Light J, Davis V, Caliskan Y, Lentine KL. The Diagnostic Yield of Genomic Sequencing-based Genetic Kidney Disease Testing in Kidney Transplant Candidates: Experience at an Urban US Transplant Center. Transplantation. 2025 Jul 1;109(7):1201-1208. doi: 10.1097/TP.0000000000005288. Epub 2025 Jan 14. PMID 39819994
- See also: Julie S. Kennan, Nephrology News & Issues, November 2022, with interview of co-PI Dr. Lentine "Black Americans with hypertension open to genetic testing, concerned about kidney disease" — https://www.healio.com/news/nephrology/20221108/black-americans-with-hypertension-open-to-genetic-testing-concerned-about-kidney-disease